CLINICAL TRIAL: NCT06571058
Title: Feasibility Testing of a Urinary Drainage Bag Securement Device to Improve Patient and Clinician Ambulation Experiences
Brief Title: B3 Buddy for Securing Urinary Drainage Bag to Patient While Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Karen Meade, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-22357; NCI-2024-04927 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-06-27; First posted 2024-08-26 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Urinary System Disorder
MeSH Terms: conditions — Urologic Diseases | interventions — Insemination, Artificial, Heterologous; Early Intervention, Educational; Educational Status; Methods; Physical Examination; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clinicians (B3 Buddy) (Experimental): Clinicians receive a short instructional session, secure the urinary drainage bag to the patient using the B3 Buddy device. Clinicians also assist patient with walking and then remove the device and return urinary drainage bag to the standard position on study.
  Interventions: Other: Assistance; Other: Educational Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Procedure: Remove
- Patients (B3 Buddy) (Experimental): Patients receive a short instructional session, wear the B3 Buddy device to secure urinary drainage bag and walk approximately 90 feet before urinary drainage bag is returned to the standard position on study.
  Interventions: Other: Educational Intervention; Device: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Walking

INTERVENTIONS:
Other: Assistance — Assist patient with walking approximately 90 feet
  Other Names: Aid; Assist; Help
  Arms: Clinicians (B3 Buddy)
Other: Educational Intervention — Receive a short instructional session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Device: Medical Device Usage and Evaluation — Wear the B3 Buddy device
  Arms: Patients (B3 Buddy)
Other: Medical Device Usage and Evaluation — Secure the urinary drainage bag to the patient using the B3 Buddy device
  Arms: Clinicians (B3 Buddy)
Other: Questionnaire Administration — Ancillary studies
Procedure: Remove — Remove the device and return urinary drainage bag to the standard position
  Other Names: Removal
  Arms: Clinicians (B3 Buddy)
Other: Walking — Walk approximately 90 feet
  Other Names: Ambulation; By Foot; On Foot; Walk
  Arms: Patients (B3 Buddy)

SUMMARY:
This clinical trial tests how well the Bag Below Bladder (B3) Buddy device works in securing urinary drainage bags while walking. Keeping a urinary drainage bag below the bladder is the standard of care to maintain urine flow and prevent urine from backing up into the bladder. Despite the use of modern urinary drainage bags for over 60 years, workarounds, including hooking the bag into pants pockets, are being used to secure the bags while walking. The B3 Buddy may help keep the urinary drainage bag at the proper level for drainage while walking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the acceptability of the B3 Buddy, from the patient's perspective.

II. To evaluate the usability of the B3 Buddy, from the clinician's perspective.

OUTLINE: Patients are assigned to 1 of 2 groups.

PATIENTS: Patients receive a short instructional session, wear the B3 Buddy device to secure urinary drainage bag and walk approximately 90 feet before urinary drainage bag is returned to the standard position on study.

CLINICIANS: Clinicians receive a short instructional session, secure the urinary drainage bag to the patient using the B3 Buddy device. Clinicians also assist patient with walking and then remove the device and return urinary drainage bag to the standard position on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT PARTICIPANT: Must be English-speaking
* PATIENT PARTICIPANT: Able to comprehend and agree to consent
* PATIENT PARTICIPANT: Able to read and complete the Acceptability of Implementation Measure (AIM) survey
* PATIENT PARTICIPANT: Be willing to participate using the B3 Buddy device
* PATIENT PARTICIPANT: Have an indwelling urinary catheter or urostomy device connected to a drainage bag
* PATIENT PARTICIPANT: Have no restrictions in ambulation
* CLINICIAN PARTICIPANT: Must be English-speaking
* CLINICIAN PARTICIPANT: Able to comprehend and agree to consent
* CLINICIAN PARTICIPANT: Able to read and complete the System Usability Scale (SUS) survey
* CLINICIAN PARTICIPANT: Be willing to participate using the B3 Buddy device
* CLINICIAN PARTICIPANT: Have a professional role in assisting patients in ambulation in normal workday activities

Exclusion Criteria:

* Those patient participants that have more than one urinary-like drainage bags will be excluded. This exclusion is due to the limited prototype samples available to the research team. Limiting one device for one patient with multiple drainage bags may not allow for accurate assessment of the B3 Buddy device

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Meade, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinicians (B3 Buddy) | Patients (B3 Buddy)
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinicians (B3 Buddy) | Patients (B3 Buddy) | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 6 | 26
  >=65 years | 0 | 15 | 15
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex demographics were not collected for the Clinicians arm
  Participants
    number analyzed (Participants) | 0 | 21 | 21
    Female |  | 6 | 6
    Male |  | 15 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 21 | 41
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Device
Description: The proportion of patients who find the device acceptable will be determined with the Acceptability of Implementation Measure tool. he AIM has 4 Likert items, ranging from 1 (for "completely disagree") to 5 (for "completely agree"). A higher number indicates greater acceptability. If a patient marked 3 or more items with at least a "4," the device was considered acceptable. The device will be considered acceptable if at least 70% of patient participants find the device acceptable, which will be calculated by survey responses.
Time Frame: Up to 17 minutes
Population: Acceptability of device was only measured for patient arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clinicians (B3 Buddy) | Patients (B3 Buddy)
Number analyzed (Participants) | 0 | 21
percentage of participants |  | 100 [83.9 to 100]

2. Primary Outcome: Usability of Device
Description: Clinicians perception of usability will be determined with the System Usability Scale. The System Usability Scale score ranges from 0 to 100, where 100 represents the highest possible perceived usability. The device will be considered usable if the overall mean score is 68 or greater, which will be calculated by survey responses.
Time Frame: Up to 20 minutes
Population: Usability of device was only measured for the clinician arm
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Clinicians (B3 Buddy) | Patients (B3 Buddy)
Number analyzed (Participants) | 20 | 0
score on a scale | 90.1 [84.9 to 95.3] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected during intervention for each participant, a time period that lasted up to 20 minutes.
Arm/Group | Clinicians (B3 Buddy) | Patients (B3 Buddy)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT06571058/Prot_SAP_003.pdf
  • Informed Consent Form: Clinician Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT06571058/ICF_001.pdf
  • Informed Consent Form: Patient Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT06571058/ICF_002.pdf